CLINICAL TRIAL: NCT05471206
Title: Evaluation of Gastrointestinal pH and Motility by Using the SmartPill® Motility Capsules After the Consumption of Milk in Symptomatic Milk Intolerant and Asymptomatic Subjects
Brief Title: Evaluation of Gastrointestinal pH and Motility After the Consumption of Milk
Acronym: ROVER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of commercialization of the medical devices
Sponsor: Lactalis (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A02653-38
Record Dates: First submitted 2022-07-11; First posted 2022-07-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk intolerant volunteers (Experimental)
  Interventions: Other: Milk and SmartPill intakes
- Milk tolerant volunteers (Active Comparator)
  Interventions: Other: Milk and SmartPill intakes

INTERVENTIONS:
Other: Milk and SmartPill intakes — During visit V2, the subject will ingest the SmartPill capsule. Then, subjects will drink milk.

SUMMARY:
This pilot study is designed as a monocentric, open label, interventional, parallel arms, controlled clinical trial. The aim of the study is to assess the gastrointestinal pH and motility after the consumption of milk.

The clinical study is categorized as an interventional research involving the human person with low risks and constraints (RIPH 2) and which does not assess a health product.

The milk and medical device used in this clinical study are both authorized and already commercialized in France.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years (limits included),
* BMI between 18.5 and 30 kg/m² (limits included),
* Able and willing to drink 250mL of milk in 5 minutes,
* Good general and mental health with in the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or clinical examination,
* Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form,
* Affiliated with a social security scheme,
* For milk intolerant subjects: self-reporting symptoms after drinking milk and drinking less than 150mL of cow's milk (lactose-free milk not included) per week (assessed by the gastrointestinal symptoms questionnaire filled out at V0).
* For milk tolerant subjects: drinking at least 700mL of cow's milk (lactose-free milk not included) per week (assessed by the gastrointestinal symptoms questionnaire filled out at V0).

Exclusion Criteria:

* Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble, uncontrolled arterial hypertension or other metabolic disorder,
* Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, arthritis, etc.) or disorders found to be inconsistent with the conduct of the study by the investigator,
* Suffering from any obstructive or restrictive respiratory syndrome (COPD, asthma, etc.) that may impact breath test measurements,
* Suffering from a gastro-intestinal pathology (inflammatory bowel disease, Crohn disease, ulcerative colitis, irritable bowel syndrome, celiac disease, gluten hypersensitivity, small intestinal bacterial overgrowth, diverticulitis, polyps, constipation, esophageal motility abnormality, history of gastric bezoar...), or other gastro-intestinal disorders found to be inconsistent with the conduct of the study by the investigator,
* Suffering from any disorder found to be inconsistent with the conduct of the study by the investigator,
* With a history of gastro-intestinal surgery (only appendectomy is accepted),
* With swallowing problems,
* With a known or suspected allergy to cows' milk protein,
* With a lactose intolerance diagnosed by a positive Lactose Breath Test,
* Pregnant or lactating women or intending to become pregnant during the study,
* Under treatment or dietary supplement which could significantly affect the gut motility and/or interfere with gastric emptying time and/or affect the gut pH during the study according to the investigator or stopped less than 15 days before the V0 visit (examples: NSAIDs, proton pump inhibitors, prokinetics, treatments against diarrhea or constipation, etc.),
* Regular intake of dietary supplements containing prebiotics, probiotics or symbiotics, or stopped less than 3 months before the V0 visit,
* With significant change in food habits or in physical activity in the 3 months before the V0 visit or not agreeing to keep them unchanged throughout the study,
* Weight loss or gain > 5% of body weight in the 6 months before the study,
* With a current diet or stopped less than 3 months before the study,
* With a current eating disorder (anorexia nervosa, bulimia, etc.) according to the investigator,
* Consuming more than 2 standard drinks of alcoholic beverage daily regularly and not agreeing to keep alcohol consumption habits unchanged throughout the study,
* Smoker (electronic cigarette not allowed),
* Consuming illicit drugs,
* Having an implanted or portable electro-mechanical medical device (such as pacemakers, defibrillators, infusion pumps…etc),
* Taking part in another clinical trial or being in the exclusion period of a previous clinical trial,
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision,
* Presenting a psychological or linguistic incapability to sign the informed consent,
* Impossible to contact in case of emergency.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this study is the AUC of pH, defined between 0 and 120 minutes after ingestion of milk, expressed in pH.min. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Guerville, Study Director — Lactalis
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No